CLINICAL TRIAL: NCT06135636
Title: Assessing Interventions to Increase Tdap Acceptance for Non-birthing Partners in Pregnancy
Acronym: ITAPP
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Laurie Griffin, Principal Investigator, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2095986
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Non-birthing Partner Vaccination in Pregnancy; Tdap - Tetanus, Diphtheria and Acellular Pertussis Vaccination; Vaccine Exposure During Pregnancy
Keywords: Tdap; Vaccine; Vaccine access; Non-birthing partner; Pregnancy
MeSH Terms: conditions — Diphtheria | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual Care (No Intervention): No up-front education, routine counseling as per their primary provider's standard practice, and written education on cocooning and recommendation for partner Tdap vaccination provided upon completion of the postpartum survey
- Upfront Education Only (Experimental): Direct verbal and written education at the time of enrollment on cocooning and recommendation for partner Tdap vaccination prior to delivery
  Interventions: Behavioral: Education
- Upfront Education and Vaccination Administration: (Experimental): Direct verbal and written education at the time of enrollment on cocooning and recommendation for partner Tdap vaccination prior to delivery plus the option to receive Tdap at their convenience at the WIH obstetric care clinic.
  Interventions: Behavioral: Education; Biological: Vaccine administration

INTERVENTIONS:
Behavioral: Education — Direct verbal and written education at the time of enrollment on cocooning and recommendation for partner Tdap vaccination prior to delivery
  Arms: Upfront Education Only; Upfront Education and Vaccination Administration:
Biological: Vaccine administration — Option to receive Tdap at their convenience at the WIH obstetric care clinic provided to participant
  Arms: Upfront Education and Vaccination Administration:

SUMMARY:
The goal of this randomized control trial is to assess if prenatal vaccine education and in-office vaccination administration for non-birthing partners of pregnant patients increases Tdap vaccination rates compared to usual care.

The main question[s] it aims to answer are:

* To assess whether compared to standard prenatal care, targeted prenatal education regarding Tdap vaccination recommendations with and without in office vaccination opportunities improves Tdap uptake among non-birthing partners of pregnant patients.
* To assess whether non-birthing partners presenting for Tdap vaccination are willing to accept dual vaccination with Tdap and influenza.

Participants will receive direct verbal and written education at the time of enrollment on cocooning and recommendation for partner Tdap vaccination prior to delivery with or without the option to receive Tdap at their convenience at the WIH obstetric care clinic.

If there is a comparison group: Researchers will compare "Upfront Education" and "Upfront Education and Vaccination Administration" to "Usual care" to see if education and/or the offer for vaccination in the office increases Tdap vaccine acceptance for non-birthing partners.

DETAILED DESCRIPTION:
Vaccination plays a critical role in decreasing the morbidity and mortality of vaccine-preventable diseases. During pregnancy, maternal vaccination increases neonatal immunity via passive immunity through antibody transmission across the placenta. However, when compared to relying on maternal vaccination alone, "cocooning"-the term for vaccinating all caregivers of newborns- is more effective in reducing neonatal morbidity and mortality from vaccine-related illnesses. Accordingly, the American College of Obstetrician and Gynecologist (ACOG) and Centers for Disease Control (CDC) both recommend that all caregivers be up-to-date on Tdap (Tetanus, Diphtheria and Pertussis), COVID-19, and influenza vaccinations to minimize risk of exposure of vaccine preventable diseases for postpartum individuals and neonates. Unfortunately, the majority of reproductive-aged individuals are not up to date on their routine vaccinations. For example, it is recommended that all adults ≥ 19 years old receive Tdap at least once in their lifetime with Td or Tdap boosters every 10 years; however, only 32.5% of reproductively aged individuals in the United States are vaccinated to TDAP.

The CDC has made calls for unique programs to minimize "missed opportunities," or when an eligible individual is at a health care encounter but fails to be vaccinated completely. Prenatal care is a time in which pregnant and non-pregnant reproductively aged individuals frequently participate in health care. Women who reported that a prenatal care provider offered vaccination in office or via referral were the most likely to receive a vaccination to influenza and Tdap compared to those who only received a vaccine recommendation or those who received no recommendation. This indicates that reducing barriers to vaccination (i.e. immediate in office vaccination), not just recommending vaccination, maximizes vaccine uptake. Prior small studies have demonstrated that the majority of parents of infants admitted to the Neonatal Intensive Care Unit and, in one small, non-randomized acceptability study, nearly two thirds of non-birthing partners accepted Tdap vaccination when offered during prenatal care. However, the majority of prenatal care providers do not offer vaccination to non-birthing partners due to administrative burden, a clear "missed opportunity" for vaccination. Programs expanding vaccine education and administration to non-birthing partners during routine prenatal care has yet to be explored, but such programs have the potential to improve perinatal and neonatal outcomes, thereby improving the health of multiple generations.

Investigators propose to implement a study of vaccine education and administration targeted specifically at Tdap vaccination for non-birthing partners of pregnant patients. The project will assess targeted educational tools for the counseling of non-birthing partners on Tdap recommendations and cocooning, as well as the impact of in-office vaccination opportunities on vaccine uptake for non-birthing partners during prenatal care.

ELIGIBILITY:
Inclusion Criteria:

1. Partners of pregnant patients who are receiving their prenatal care at the OGCC
2. 19-50 years old: This age range was selected as 19 years is both the age at which adult Tdap vaccination is recommended by the CDC as well as the age for the State supplied adult Tdap and Influenza Vaccines. Fifty years old is the upper limit of "reproductively aged individuals, the target population for this study.
3. Have not or are unsure if they have received the adult Tdap vaccine or booster in the last 10 years: In addition to the CDC recommendation for adult Tdap vaccination and Td or Tdap booster every 10 years, the CDC recommends vaccination for any adult who is unsure of their vaccination status to ensure they are vaccinated as repeat vaccination does not cause additional harm.
4. Fluency in English or Spanish: Consents, surveys, and Tdap and cocooning information will be available in both languages.

Exclusion Criteria:

1. Latex allergy: Contraindication to the state supplied Tdap vaccine
2. Lethal fetal anomaly diagnosed prior to enrollment to prevent undue distress with follow-up postpartum

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Tdap vaccination rate for non-birthing partners | During pregnancy though 1 week postpartum
  To assess whether compared to standard prenatal care, targeted prenatal education regarding Tdap vaccination recommendations with and without in office vaccination opportunities improves Tdap uptake among non-birthing partners of pregnant patients.

SECONDARY OUTCOMES:
Dual vaccination rates for non-birthing partners | During pregnancy though 1 week postpartum
  To assess whether non-birthing partners presenting for Tdap vaccination are willing to accept dual vaccination with Tdap and influenza.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Griffin, MD/PhD, Principal Investigator — Women and Infants Hospital
Locations (1):
- Women and Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
Data collected in this study will not be shared with other researchers.